CLINICAL TRIAL: NCT04344119
Title: Assessment of Skin Manifestations Occuring During Covid-19 Infection With a Special Focus on Chilbains
Brief Title: Assessment of Chilbains Occuring During Covid-19 Infection
Acronym: ChilblainCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20dermatocovid01
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-04

CONDITIONS: Skin Manifestations; COVID; Chilblains
MeSH Terms: conditions — Skin Manifestations; Chilblains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, skin biopsy, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Some patients infected by covid-19 develop skin manifestations. These manifestations are still not well known and there pathophysiology remain unclear. Among them, acral manifestation resembling to chilblains appears frequent and quite specific. The aim of this project is to better characterize the cutaneous manifestations occurring during Covid-19 infection with a special focus on chilblains. These acral manifestation could be due to a direct viral effect, but also to microthrombosis or vascularitis. Understanding the pathomechanisms involved could provide interesting clue for understanding not only the skin manifestations but also some of the other systemic symptoms associated to covid-19 infection. This study plan to characterize these acral manifestations by analyzing the clinical and dermoscopic patterns and to correlate them with the non-invasive vascular explorations but also immune and coagulopathy explorations that are done in the CHU of Nice in covid-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients with proven covid infection (using PCR, serum antibody or lung TDM) and presenting at least one cutaneous lesions that occurred during the infection.

Max Age: 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients with covid infection presenting with skin manifestations
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-04-09 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinical skin manifestations | 3 months
  Type and description of the skin manifestations with a special focus on patients with chilblains

SECONDARY OUTCOMES:
Histology and biological data | 3 months
  Data on Histology (HE staining and immunofluorescence) and on biology (blood cells counts, CRP and immune profile) will be collected in covid patient with skin manifestation
Non invasive vascular examination | 3 months
  Vascular examination will be performed by Capillaroscopy, laser-doppler or lung TDM if clinically required

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

REFERENCES:
- [Derived] Hubiche T, Cardot-Leccia N, Le Duff F, Seitz-Polski B, Giordana P, Chiaverini C, Giordanengo V, Gonfrier G, Raimondi V, Bausset O, Adjtoutah Z, Garnier M, Burel-Vandenbos F, Dadone-Montaudie B, Fassbender V, Palladini A, Courjon J, Mondain V, Contenti J, Dellamonica J, Leftheriotis G, Passeron T. Clinical, Laboratory, and Interferon-Alpha Response Characteristics of Patients With Chilblain-like Lesions During the COVID-19 Pandemic. JAMA Dermatol. 2021 Feb 1;157(2):202-206. doi: 10.1001/jamadermatol.2020.4324. PMID 33237291